CLINICAL TRIAL: NCT06703125
Title: The Alama Project: Autism Outcomes and Neurobehavioral Markers in Young Children Born to Mothers With HIV in Kenya
Acronym: Alama
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Rebecca McNally Keehn, Assistant Professor of Pediatrics, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23171; 1R01HD116441-01 (NIH)
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Autism
Keywords: Autism; HIV; Eye tracker
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Children Undergoing Developmental Evaluation for Autism (Experimental): Young children (ages 24-72 month) who are HIV exposed but uninfected (CHEU) and young children who are HIV unexposed but uninfected (CHUU) undergoing a standard of care developmental evaluation will be enrolled into the study. After the completion of the developmental evaluation, research participation includes a one-time eye-tracking activity in which the child will view a series of different pictures and movies while their eye movements and pupil diameter are tracked and recorded.
  Interventions: Diagnostic Test: Eyelink Portable Duo

INTERVENTIONS:
Diagnostic Test: Eyelink Portable Duo — Eye-tracking data will be collected using a commercially-available remote eye-tracking system (Eyelink Portable Duo). Eye movements and pupil diameter will be collected while participants view a series of developmentally appropriate pictures and movies. The eye-tracker consists of two cameras; one that monitors eye movements and a second scene camera that monitors head movements, which permits eye tracking to take place without any equipment touching the child. Children will be asked to sit in highchair or on their the lap of the caregiver and will face a computer monitor. After a sticker is applied to the forehead of the child and brief eye-movement calibration completed, next visual stimuli (i.e., pictures and videos) will be presented on a laptop computer monitor that is placed at approximately 60-80cm from the child. The eye tracking portion of the visit will last approximately 15 minutes or until the child is no longer able to attend to pictures/videos.

SUMMARY:
The study will use a non-invasive remote eye-tracking system (Eyelink Portable Duo) to acquire a short series of eye-tracking measures to determine whether these can predict autism diagnoses in both children exposed to HIV and uninfected (CHEU) and children not exposed to HIV and uninfected (CHUU).

DETAILED DESCRIPTION:
The study will use a non-invasive remote eye-tracking system (Eyelink Portable Duo) to acquire a short series (less than 15 mins) of eye-tracking measures (e.g., looking time, pupil diameter, oculomotor dynamics), which may be associated with autism outcomes. Investigators will recruit children enrolled in the Tabiri study during or following their 24-month visit.

The Tabiri study is comparing neurodevelopmental (ND) outcomes between 24-month-old CHEU and CHUU.

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled in the Tabiri study (R01HD104552)
* CHEU or CHUU
* Children ages 24-72 months
* Caregivers of children must speak Kiswahili (local language) or English.

Exclusion Criteria:

* There will be no specific exclusion criteria. We anticipate that a small number of CHEU and CHUU will develop HIV prior to enrollment in the current study; these children will be included and will follow all general study procedures.

Ages: 24 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 850 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Agreement between eye-tracking biomarker score and autism diagnosis | Day 1
  The composite eye-tracking biomarker score, a consolidated measure based on eye-tracking indices that predict autism outcome, will be compared to the categorical autism diagnosis (autism presence/absence). Clinical diagnosis is obtained based upon a standard clinical evaluation. The evaluation will include 1) a semi-structured caregiver(s) clinical interview to gather information about developmental history and autism symptoms and 2) a battery of standardized child clinical observational measures. The evaluation will be conducted over a one-time 2- to 3-hour clinical autism evaluation. Eye-tracking will be recorded immediately following the clinical evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca McNally Keehn, Principal Investigator — IU School of Medicine
Locations (1):
- Moi Teaching and Referral Hospital, Eldoret, Kenya, Kenya

IPD SHARING:
Plan to Share IPD: No